CLINICAL TRIAL: NCT03080207
Title: Comparison of Efficacy of Platelets / Platelet Enriched Plasma Regard (PRP) Method, Complex Decongestive Physiotherapy and Low Level Laser in Treatment of Lower Extremity Lymphoedema
Brief Title: Platelet Rich Plasma, Complex Decongestive Physiotherapy and Low Level Laser in Treatment of Lower Extremity Lymphoedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Akgul, Prof.Dr., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSA-2017-22398
Record Dates: First submitted 2017-03-05; First posted 2017-03-15 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Lower Extremity Lymphedema
Keywords: Lower Extremity Lymphedema; Physiotherapy; Complex Decongestive Physiotherapy; Low Level Laser; Platelet rich plasma
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Platelets / Platelet Enriched Plasma Regard (PRP) Method (Experimental)
  Interventions: Procedure: PRP method
- Complex Decongestive Physiotherapy (Experimental)
  Interventions: Procedure: Low Level Laser
- Low Level Laser (Experimental)
  Interventions: Procedure: Complex Decongestive Physiotherapy

INTERVENTIONS:
Procedure: PRP method — It will first be placed on a 25 cc venous blood centrifuge in anticoagulated tubes containing acid citrate dextrose (ACD), and autologous venous blood will be centrifuged at 3200 rpm for 15 minutes. Using the PRP kit, the plasma rich in platelet volume of about 3 cc volume will be removed. This will be activated by the addition of platelet agonists such as thrombin, calcium gluconate or calcium chloride. Injections should be administered subcutaneously for 2-3 weeks, 3-4 times for inguinal, popliteal region and ankle for a total of 12 weeks. Also, all patients in this groups have received Complex Decongestive Physiotherapy (Manual lymph drainage (MLD), skin care, compression therapy and active therapeutic exercise).
  Arms: Platelets / Platelet Enriched Plasma Regard (PRP) Method
Procedure: Low Level Laser — Low Density Laser treatment will be applied for the first 4 weeks every 12 weeks, the remaining 8 weeks 2 days / week. A total of 9 regions (6 point inguinal region and 3 points popliteal region) are to be applied by applying the laser head close to the skin (20000 Hz, 1.5 J / cm2) with the laser device and the regions where lymph nodes and lymph pathways are dense.
  During the application, the patient will be in the supine position for the popliteal region, with the patient in the supine position for the inguinal region and the legs free in the abdomen.Also, all patients in this groups have received Complex Decongestive Physiotherapy (Manual lymph drainage (MLD), skin care, compression therapy and active therapeutic exercise).
  Arms: Complex Decongestive Physiotherapy
Procedure: Complex Decongestive Physiotherapy — Complex Decongestive Physiotherapy (CDP) consists of four basic components and two phases. Four basic components; Manual lymph drainage (MLD), skin care, compression therapy and therapeutic exercise. Phase I (intense phase): It is also referred to as the phase of reducing the remission. In this phase, skin care and compression bandages are renewed after daily MLD application. The patient is taught how to bandage on his own. (Phase I, 4 weeks) The duration of phase I may vary according to the patient. In Phase II, MLD can be administered 2 or 3 times per week depending on the needs of the individual. In this case, the patient is followed by home program. Our cases will be treated in Phase I every day for 12 weeks in total and 2 days / week in Phase II according to KBF phases. All patients in this group have received only Complex Decongestive Physiotherapy.
  Arms: Low Level Laser

SUMMARY:
At the end of the study, comparative information about the effects of PRP, complex decongestive physiotherapy and low level laser on edema volume, range of motion, muscle strength, functional capacity and quality of life will be obtained in the treatment of patients with lower limb lymphedema.

Since there is no study about this field in the literature, this study will provide new and valuable contributions about treatment of lower extremity lymphedema for the researchers and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Having lower extremity lymphedema
* To be older than 18 ages.

Exclusion Criteria:

* Having received radiotherapy treatment in the last 6 months,
* Having received physiotherapy treatment in the last 6 months,
* General health status is not eligible for treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 12 weeks

SECONDARY OUTCOMES:
Lower-extremity-circumference | 12 weeks
Numeric rating scale | 12 weeks
6 minutes walking test | 12 weeks
Tissue dielectric constant Questionnaire | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Akgul, Prof.Dr., Principal Investigator — Istanbul University; Ela Tarakci, Assoc.Dr., Study Director — Istanbul University; Nilay Arman, PhD, PT, Study Director — Istanbul University; Tugba Civi, PT, Study Director — Istanbul University; Musa Cirak, MD, DR, Study Director — Bakirkoy Dr.Sadi Konuk Education and Research Hospital
Locations (1):
- Istanbul University Faculty of Health Science, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akgul A, Tarakci E, Arman N, Civi T, Irmak S. A Randomized Controlled Trial Comparing Platelet-Rich Plasma, Low-Level Laser Therapy, and Complex Decongestive Physiotherapy in Patients with Lower Limb Lymphedema. Lymphat Res Biol. 2020 Oct;18(5):439-447. doi: 10.1089/lrb.2019.0064. Epub 2020 Feb 19. PMID 32073990